CLINICAL TRIAL: NCT02621281
Title: Clinical Impact of Hypothermic Machine Perfusion in Renal Transplant Recipients
Acronym: CIHMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: The First Hospital of Jilin University (Other); 303rd Hospital of the People's Liberation Army (Other); Fuzhou General Hospital (Other)
Responsible Party: Principal Investigator, Ding,Chenguang, PHD, First Affiliated Hospital Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LPT-G-1501
Record Dates: First submitted 2015-11-29; First posted 2015-12-03 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Delayed Function of Renal Transplant
Keywords: hypothermic machine perfusion; Kidney Transplantation; Delayed graft function; perfusion pressure
MeSH Terms: conditions — Delayed Graft Function | interventions — Cryopreservation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cold storage (Active Comparator): In this randomized clinical trial, 200 kidney pairs from deceased donors will be included in the study, which will be randomly assigned, one kidney to machine perfusion and the other to cold storage. In machine perfusion group, patients will be analyzed by two subgroups based on pressure, resistance index and perfusion time duration.
  Interventions: Device: cold storage
- Kidney Transporter machines (Active Comparator): In this randomized clinical trial, 200 kidney pairs from deceased donors will be included in the study, which will be randomly assigned, one kidney to machine perfusion and the other to cold storage. In machine perfusion group, patients will be analyzed by two subgroups based on pressure, resistance index and perfusion time duration.
  Interventions: Device: Kidney Transporter machines

INTERVENTIONS:
Device: Kidney Transporter machines — Kidney Transporter gently pumps the special cold solution through the kidney which outside the body.
  Arms: Kidney Transporter machines
Device: cold storage — The kidneys procurement from the donor will be cold stored using some cold preservation solution.
  Arms: cold storage

SUMMARY:
This is a multi-centers prospective, randomized, controlled trial. This trial will investigate the clinical outcome of kidney transplant recipients whose kidneys are under two different forms of organ preservation--hypothermic machine perfusion vs. static cold storage. Factors during the machine perfusion, such as the pressure, flow rate, and resistance index will also be investigated.

DETAILED DESCRIPTION:
In this randomized clinical trial, 200 kidney pairs from deceased donors will be included in the study, which will be randomly assigned, one kidney to machine perfusion and the other to cold storage. All 400 patients will be followed for 1 year. The primary endpoint is delayed graft function (requiring dialysis in the first week after transplantation) and duration of delayed graft function. The second endpoints: GFR at week 1, month3, month6 and month 12 post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Donor

  1. Comply with the national DCD（donor after citizen death) guideline
  2. No high risk activities: such as history of drug abuse, history of intravenous drug use and risky sexual behavior
  3. No malignant melanoma, metastatic cancer, or incurable cancer; some of the early stages of cancer after a successful treatment can also be considered
  4. No active, untreated systemic bacterial, viral or fungal infection;
  5. Patients definitely identified
  6. Mechanical perfusion RI (resistance index ) [0.18, 0.50]

Recipient:

1. Age> = 16 years old, male or female
2. BMI<28
3. First Renal transplantation
4. Not in pregnancy or lactation, pregnancy test was negative, and promise not to be pregnant during treatment.
5. Before the clinical trial, Patient sign informed consent voluntarily

Exclusion Criteria:

* Donor

  1. Older than 50 years old
  2. Serum HBV (hepatitis B virus), HCV (hepatitis C virus), HIV positive
  3. Donor kidney cold storage time over 30 hours
  4. Warm ischemia time over 20 minutes
  5. Other reagents are added perfusion for regulation of donor renal function

Recipient:

1. Double organ or multi-organ transplant
2. Blood type-incompatible
3. Patients with other malignant diseases

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
The rate of Delayed graft function | the first week after transplant
  Delayed graft function (DGF) is a common complication of renal transplantation. DGF can be diagnosed according to the three aspects below.
  i. Need for postoperative dialysis: Need for dialysis in the first week after transplant once hyperacute rejection, vascular and urinary tract complications and hyperkalemia are ruled out.
  ii. Urine output and serum creatinine: 1) Rise in serum Cr at 6-8 h post-operatively or <300 ml of urine despite adequate volume and diuretics. 2) Urine output <1 L in 24 h and <25% fall in serum creatinine from baseline in first 24 h post-transplant. 3) Urine output <75 mL/h in first 48 h or failure of serum Cr to decrease by 10% in the first 48 h. 4) Serum creatinine increases or remains unchanged or decreases <10%/day during 3 consecutive days postoperatively. 5) Serum creatinine >2.5mg/dL on Day 7 or need for post-transplant hemodialysis.6) Time required for the kidney to reach CrCl>10 mL/min greater than 1 week.

SECONDARY OUTCOMES:
Estimated Glomerular Filtration Rate | 1 week, three months, six months, 12 months after kidney transplant
  Glomerular filtration rate (GFR) is the volume of fluid filtered from the renal (kidney) glomerular capillaries into the Bowman's capsule per unit time.[3] Central to the physiologic maintenance of GFR is the differential basal tone of the afferent and efferent arterioles (see diagram). In other words, the filtration rate is dependent on the difference between the higher blood pressure created by vasoconstriction of the input or afferent arteriole versus the lower blood pressure created lesser vasoconstriction of the output or efferent arteriole.

CONTACTS AND LOCATIONS:
Overall Officials: Wujun Xue, PhD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital Xi'an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Result] Moers C, Smits JM, Maathuis MH, Treckmann J, van Gelder F, Napieralski BP, van Kasterop-Kutz M, van der Heide JJ, Squifflet JP, van Heurn E, Kirste GR, Rahmel A, Leuvenink HG, Paul A, Pirenne J, Ploeg RJ. Machine perfusion or cold storage in deceased-donor kidney transplantation. N Engl J Med. 2009 Jan 1;360(1):7-19. doi: 10.1056/NEJMoa0802289. PMID 19118301
- [Result] Moers C, Pirenne J, Paul A, Ploeg RJ; Machine Preservation Trial Study Group. Machine perfusion or cold storage in deceased-donor kidney transplantation. N Engl J Med. 2012 Feb 23;366(8):770-1. doi: 10.1056/NEJMc1111038. No abstract available. PMID 22356343
- [Result] Tapiawala SN, Tinckam KJ, Cardella CJ, Schiff J, Cattran DC, Cole EH, Kim SJ. Delayed graft function and the risk for death with a functioning graft. J Am Soc Nephrol. 2010 Jan;21(1):153-61. doi: 10.1681/ASN.2009040412. Epub 2009 Oct 29. PMID 19875806
- [Result] Perico N, Cattaneo D, Sayegh MH, Remuzzi G. Delayed graft function in kidney transplantation. Lancet. 2004 Nov 13-19;364(9447):1814-27. doi: 10.1016/S0140-6736(04)17406-0. PMID 15541456
- [Result] Yarlagadda SG, Coca SG, Formica RN Jr, Poggio ED, Parikh CR. Association between delayed graft function and allograft and patient survival: a systematic review and meta-analysis. Nephrol Dial Transplant. 2009 Mar;24(3):1039-47. doi: 10.1093/ndt/gfn667. Epub 2008 Dec 22. PMID 19103734
- [Result] Jochmans I, Moers C, Smits JM, Leuvenink HG, Treckmann J, Paul A, Rahmel A, Squifflet JP, van Heurn E, Monbaliu D, Ploeg RJ, Pirenne J. Machine perfusion versus cold storage for the preservation of kidneys donated after cardiac death: a multicenter, randomized, controlled trial. Ann Surg. 2010 Nov;252(5):756-64. doi: 10.1097/SLA.0b013e3181ffc256. PMID 21037431
- [Result] Treckmann J, Moers C, Smits JM, Gallinat A, Maathuis MH, van Kasterop-Kutz M, Jochmans I, Homan van der Heide JJ, Squifflet JP, van Heurn E, Kirste GR, Rahmel A, Leuvenink HG, Pirenne J, Ploeg RJ, Paul A. Machine perfusion versus cold storage for preservation of kidneys from expanded criteria donors after brain death. Transpl Int. 2011 Jun;24(6):548-54. doi: 10.1111/j.1432-2277.2011.01232.x. Epub 2011 Feb 17. PMID 21332580
- [Result] Patel SK, Pankewycz OG, Nader ND, Zachariah M, Kohli R, Laftavi MR. Prognostic utility of hypothermic machine perfusion in deceased donor renal transplantation. Transplant Proc. 2012 Sep;44(7):2207-12. doi: 10.1016/j.transproceed.2012.07.129. PMID 22974956
- [Result] Jochmans I, Moers C, Smits JM, Leuvenink HG, Treckmann J, Paul A, Rahmel A, Squifflet JP, van Heurn E, Monbaliu D, Ploeg RJ, Pirenne J. The prognostic value of renal resistance during hypothermic machine perfusion of deceased donor kidneys. Am J Transplant. 2011 Oct;11(10):2214-20. doi: 10.1111/j.1600-6143.2011.03685.x. Epub 2011 Aug 11. PMID 21834917
- [Result] Doorschodt BM, Schreinemachers MC, Behbahani M, Florquin S, Weis J, Staat M, Tolba RH. Hypothermic machine perfusion of kidney grafts: which pressure is preferred? Ann Biomed Eng. 2011 Mar;39(3):1051-9. doi: 10.1007/s10439-010-0228-7. Epub 2010 Dec 16. PMID 21161683
- [Result] Patel SK, Pankewycz OG, Weber-Shrikant E, Zachariah M, Kohli R, Nader ND, Laftavi MR. Effect of increased pressure during pulsatile pump perfusion of deceased donor kidneys in transplantation. Transplant Proc. 2012 Sep;44(7):2202-6. doi: 10.1016/j.transproceed.2012.07.109. PMID 22974955
- [Result] Sung RS, Christensen LL, Leichtman AB, Greenstein SM, Distant DA, Wynn JJ, Stegall MD, Delmonico FL, Port FK. Determinants of discard of expanded criteria donor kidneys: impact of biopsy and machine perfusion. Am J Transplant. 2008 Apr;8(4):783-92. doi: 10.1111/j.1600-6143.2008.02157.x. Epub 2008 Feb 19. PMID 18294347
- [Result] Cantafio AW, Dick AA, Halldorson JB, Bakthavatsalam R, Reyes JD, Perkins JD. Risk stratification of kidneys from donation after cardiac death donors and the utility of machine perfusion. Clin Transplant. 2011 Sep-Oct;25(5):E530-40. doi: 10.1111/j.1399-0012.2011.01477.x. Epub 2011 May 18. PMID 21585547
- [Result] Akoh JA. Kidney donation after cardiac death. World J Nephrol. 2012 Jun 6;1(3):79-91. doi: 10.5527/wjn.v1.i3.79. PMID 24175245
- [Result] Chapal M, Le Borgne F, Legendre C, Kreis H, Mourad G, Garrigue V, Morelon E, Buron F, Rostaing L, Kamar N, Kessler M, Ladriere M, Soulillou JP, Launay K, Daguin P, Offredo L, Giral M, Foucher Y. A useful scoring system for the prediction and management of delayed graft function following kidney transplantation from cadaveric donors. Kidney Int. 2014 Dec;86(6):1130-9. doi: 10.1038/ki.2014.188. Epub 2014 Jun 4. PMID 24897036
- [Result] Irish WD, Ilsley JN, Schnitzler MA, Feng S, Brennan DC. A risk prediction model for delayed graft function in the current era of deceased donor renal transplantation. Am J Transplant. 2010 Oct;10(10):2279-86. doi: 10.1111/j.1600-6143.2010.03179.x. PMID 20883559
- [Result] Jeldres C, Cardinal H, Duclos A, Shariat SF, Suardi N, Capitanio U, Hebert MJ, Karakiewicz PI. Prediction of delayed graft function after renal transplantation. Can Urol Assoc J. 2009 Oct;3(5):377-82. doi: 10.5489/cuaj.1147. PMID 19829730
- [Derived] Tingle SJ, Thompson ER, Figueiredo RS, Moir JA, Goodfellow M, Talbot D, Wilson CH. Normothermic and hypothermic machine perfusion preservation versus static cold storage for deceased donor kidney transplantation. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD011671. doi: 10.1002/14651858.CD011671.pub3. PMID 38979743